CLINICAL TRIAL: NCT05948332
Title: Definition and Management of Right Ventricular Injury in Adult Patients Receiving Extracorporeal Membrane Oxygenation for Respiratory Support Using the Delphi Method: A PRORVnet - Expert Consensus Statements
Brief Title: Definition and Management of Right Ventricular Injury in Adult Patients Receiving Extracorporeal Membrane Oxygenation
Status: Completed | Type: Observational
Sponsor: Prashant Nasa (Other)
Responsible Party: Sponsor-Investigator, Prashant Nasa, HOD, Critical Care Medicine, NMC Specialty Hospital
Organization: NMC Specialty Hospital (Other)
Other Study IDs: RVI_ECMO
Record Dates: First submitted 2023-07-08; First posted 2023-07-17 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Extracorporeal Circulation; Complications; Extracorporeal Membrane Oxygenation Complication; Right Heart Failure; Right Ventricular Dysfunction; Respiratory Failure; Respiratory Distress Syndrome
Keywords: Extracorporeal Membrane Oxygenation; Heart Failure; Right Ventricular Injury; Respiratory Distress Syndrome
MeSH Terms: conditions — Heart Failure; Ventricular Dysfunction, Right; Respiratory Insufficiency; Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Delphi Rounds to generate consensus opinions among Experts — The Investigators (Steering Committee) will select the experts from across the globe based on pre-specified qualification criteria and will conduct iterative Delphi rounds to generate consensus on the definition and management of acute RVI in patients with receiving V-V ECMO, among the Experts. The selection criteria will be self-assessed through a survey among the potential Experts.

SUMMARY:
The aim of this study is to identify existing definitions and therapeutic approaches for acute right ventricular injury (RVI) in patients receiving extracorporeal membrane oxygenation (ECMO) for respiratory support. The objective of the study is to generate expert consensus statements on the definition and management of acute RVI in this high-risk patient population, using a Delphi method. The standardised RVI definition during ECMO for respiratory support and a consensus-based management approach to RVI will facilitate systematic aggregation of data across clinical trials to harmonise patient selection and compare therapeutic interventions.

DETAILED DESCRIPTION:
Extracorporeal membrane oxygenation (ECMO) is increasingly being used as part of the algorithm for the management of patients with respiratory failure in whom conventional ventilatory strategies have failed to preserve gas exchange without use of settings that may result in ventilator-induced lung injury. ECMO for respiratory support may be required in critically ill patients with any of the following types of respiratory failure: a) acute respiratory distress syndrome (ARDS) of any aetiology (infectious or non-infectious, pulmonary or extrapulmonary), defined according to the Berlin criteria of ARDS, or the more recently proposed Kigali modification and the New Global definition of ARDS; b) acute reversible hypoxemic and/or hypercapnic respiratory failure of any infectious or non-infectious aetiology (including pulmonary embolism and primary graft failure in lung transplantation recipients); and c) chronic hypoxemic and/or hypercapnic respiratory failure, as a bridge to lung transplantation strategy. Right ventricular injury (RVI) may develop in the context of any of the aforementioned types of respiratory failure and is characterised by a spectrum of abnormal RV biomechanics which all have been linked to mortality. One of the main mechanisms of RVI in patients with respiratory failure is pulmonary vasoconstriction caused by hypoxaemia and/or hypercapnic acidaemia leading to elevated RV afterload. Respiratory ECMO supports or replaces pulmonary gas exchange and theoretically may reverse the aforementioned mechanism of RVI and unloads the RV. However, RVI may persist or worsen despite application of ECMO and is strongly associated with significant mortality.

There is currently no universally accepted definition for RVI in patients receiving ECMO for respiratory support or evidence-based RV-targeted therapies. This may result in underdiagnosis of this clinical entity and clinical practice variations and hence there is a need to standardise diagnostic criteria as well as clarify therapeutic management. The objective of the current investigation is to generate consensus statements by experts on the definition and management of RVI in adult patients receiving ECMO for respiratory support, using a Delphi process.

The Delphi process is a well-known mechanism for generating consensus on a specific topic by tapping into the "collective intelligence" of the panel members. The Steering Committee members conduct iterative Delphi rounds to obtain an agreement among the Experts after completing a literature search on the currently available evidence and preparing the opening statements. The members of the Steering Committee will not take part in the Delphi surveys.

The investigators will be using a modified Delphi-based methodology involving global experts from different disciplines (intensive care medicine, anaesthesia, cardiac surgery, cardiology, or a combination of two or more specialties) who meet pre-specified qualification criteria. A survey will be sent to all potential panel members prior to commencement of the Delphi rounds, to ascertain expertise in the field. The entire study will be conducted through approximately three or four rounds of Google Forms-based Delphi questionnaires. The Experts will provide opinion on the problem areas; definition and management of acute RVI in patients receiving ECMO for respiratory support. The survey is organised into three domains: Definition, RVI severity, Management strategies, and Research Priorities. The problem areas, domains and statements were generated by systematic literature review. Most of these statements require a 7-point Likert scale rating or selecting appropriate options in multiple-choice questions (MCQs). In round one, there is an option to collect feedback from participating Experts in the offered open area, which will be evaluated before the round two questionnaire. Rounds are repeated until consensus (or stable dissensus) is reached (≥70% for the Likert scale and ≥80% for MCQs). Experts will be presented with the summary results of each round, and the survey procedure will be repeated with the amended questionnaire. The Delphi rounds will continue until the required consensus (or lack thereof) and statement stability is obtained.

ELIGIBILITY:
Inclusion Criteria:

1. Working in an active Extracorporeal Life Support Organisation (ELSO) member centre for > 5 years, or clinical experience in cardiorespiratory failure for > 5 years.
2. Original research in the field of ECMO or Cardiorespiratory failure (at least one peer-reviewed publication as a leading author).

Exclusion Criteria:

People who do not meet inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Healthcare professionals involved in the management adult patients receiving Extracorporeal Membrane Oxygenation.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-11-26 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Consensus statements | Through study completion, an average of 6 months
  Consensus amongst the expert panel regarding RVI definition and management will be achieved using Delphi method which includes iterative rounds of questions; Consensus will be considered reached when a statement achieves >80% of votes for multiple-choice questions and >70% for Likert-scale statements

CONTACTS AND LOCATIONS:
Overall Officials: Vasileios Zochios, MRCP FFICM, Principal Investigator — University Hospitals of Leicester NHS Trust, Glenfied Hospital
Locations (1):
- NMC Specialty Hospital, Al Nahda, Dubai, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No
Individual participant data will be kept anonymous and be shared after the Delphi process during the publication.

REFERENCES:
- [Background] Nasa P, Azoulay E, Chakrabarti A, Divatia JV, Jain R, Rodrigues C, Rosenthal VD, Alhazzani W, Arabi YM, Bakker J, Bassetti M, De Waele J, Dimopoulos G, Du B, Einav S, Evans L, Finfer S, Guerin C, Hammond NE, Jaber S, Kleinpell RM, Koh Y, Kollef M, Levy MM, Machado FR, Mancebo J, Martin-Loeches I, Mer M, Niederman MS, Pelosi P, Perner A, Peter JV, Phua J, Piquilloud L, Pletz MW, Rhodes A, Schultz MJ, Singer M, Timsit JF, Venkatesh B, Vincent JL, Welte T, Myatra SN. Infection control in the intensive care unit: expert consensus statements for SARS-CoV-2 using a Delphi method. Lancet Infect Dis. 2022 Mar;22(3):e74-e87. doi: 10.1016/S1473-3099(21)00626-5. Epub 2021 Nov 10. PMID 34774188
- [Background] Brodie D, Slutsky AS, Combes A. Extracorporeal Life Support for Adults With Respiratory Failure and Related Indications: A Review. JAMA. 2019 Aug 13;322(6):557-568. doi: 10.1001/jama.2019.9302. PMID 31408142
- [Background] Supady A, Combes A, Barbaro RP, Camporota L, Diaz R, Fan E, Giani M, Hodgson C, Hough CL, Karagiannidis C, Kochanek M, Rabie AA, Riera J, Slutsky AS, Brodie D. Respiratory indications for ECMO: focus on COVID-19. Intensive Care Med. 2022 Oct;48(10):1326-1337. doi: 10.1007/s00134-022-06815-w. Epub 2022 Aug 9. PMID 35945343
- [Background] ARDS Definition Task Force; Ranieri VM, Rubenfeld GD, Thompson BT, Ferguson ND, Caldwell E, Fan E, Camporota L, Slutsky AS. Acute respiratory distress syndrome: the Berlin Definition. JAMA. 2012 Jun 20;307(23):2526-33. doi: 10.1001/jama.2012.5669. PMID 22797452
- [Background] Grasselli G, Calfee CS, Camporota L, Poole D, Amato MBP, Antonelli M, Arabi YM, Baroncelli F, Beitler JR, Bellani G, Bellingan G, Blackwood B, Bos LDJ, Brochard L, Brodie D, Burns KEA, Combes A, D'Arrigo S, De Backer D, Demoule A, Einav S, Fan E, Ferguson ND, Frat JP, Gattinoni L, Guerin C, Herridge MS, Hodgson C, Hough CL, Jaber S, Juffermans NP, Karagiannidis C, Kesecioglu J, Kwizera A, Laffey JG, Mancebo J, Matthay MA, McAuley DF, Mercat A, Meyer NJ, Moss M, Munshi L, Myatra SN, Ng Gong M, Papazian L, Patel BK, Pellegrini M, Perner A, Pesenti A, Piquilloud L, Qiu H, Ranieri MV, Riviello E, Slutsky AS, Stapleton RD, Summers C, Thompson TB, Valente Barbas CS, Villar J, Ware LB, Weiss B, Zampieri FG, Azoulay E, Cecconi M; European Society of Intensive Care Medicine Taskforce on ARDS. ESICM guidelines on acute respiratory distress syndrome: definition, phenotyping and respiratory support strategies. Intensive Care Med. 2023 Jul;49(7):727-759. doi: 10.1007/s00134-023-07050-7. Epub 2023 Jun 16. PMID 37326646
- [Background] Riviello ED, Kiviri W, Twagirumugabe T, Mueller A, Banner-Goodspeed VM, Officer L, Novack V, Mutumwinka M, Talmor DS, Fowler RA. Hospital Incidence and Outcomes of the Acute Respiratory Distress Syndrome Using the Kigali Modification of the Berlin Definition. Am J Respir Crit Care Med. 2016 Jan 1;193(1):52-9. doi: 10.1164/rccm.201503-0584OC. PMID 26352116
- [Background] Matthay MA, Thompson BT, Ware LB. The Berlin definition of acute respiratory distress syndrome: should patients receiving high-flow nasal oxygen be included? Lancet Respir Med. 2021 Aug;9(8):933-936. doi: 10.1016/S2213-2600(21)00105-3. Epub 2021 Apr 27. PMID 33915103
- [Background] Sato R, Dugar S, Cheungpasitporn W, Schleicher M, Collier P, Vallabhajosyula S, Duggal A. The impact of right ventricular injury on the mortality in patients with acute respiratory distress syndrome: a systematic review and meta-analysis. Crit Care. 2021 May 21;25(1):172. doi: 10.1186/s13054-021-03591-9. PMID 34020703
- [Background] Zochios V, Yusuff H, Schmidt M; Protecting the Right Ventricle Network (PRORVnet). Acute right ventricular injury phenotyping in ARDS. Intensive Care Med. 2023 Jan;49(1):99-102. doi: 10.1007/s00134-022-06904-w. Epub 2022 Oct 11. No abstract available. PMID 36219228
- [Background] Huang S, Vignon P, Mekontso-Dessap A, Tran S, Prat G, Chew M, Balik M, Sanfilippo F, Banauch G, Clau-Terre F, Morelli A, De Backer D, Cholley B, Slama M, Charron C, Goudelin M, Bagate F, Bailly P, Blixt PJ, Masi P, Evrard B, Orde S, Mayo P, McLean AS, Vieillard-Baron A; ECHO-COVID research group. Echocardiography findings in COVID-19 patients admitted to intensive care units: a multi-national observational study (the ECHO-COVID study). Intensive Care Med. 2022 Jun;48(6):667-678. doi: 10.1007/s00134-022-06685-2. Epub 2022 Apr 21. PMID 35445822
- [Background] Vieillard-Baron A, Naeije R, Haddad F, Bogaard HJ, Bull TM, Fletcher N, Lahm T, Magder S, Orde S, Schmidt G, Pinsky MR. Diagnostic workup, etiologies and management of acute right ventricle failure : A state-of-the-art paper. Intensive Care Med. 2018 Jun;44(6):774-790. doi: 10.1007/s00134-018-5172-2. Epub 2018 May 9. PMID 29744563
- [Background] Vonk Noordegraaf A, Westerhof BE, Westerhof N. The Relationship Between the Right Ventricle and its Load in Pulmonary Hypertension. J Am Coll Cardiol. 2017 Jan 17;69(2):236-243. doi: 10.1016/j.jacc.2016.10.047. PMID 28081831
- [Background] Chad T, Yusuff H, Zochios V, Pettenuzzo T, Fan E, Schmidt M; Protecting the Right Ventricle network (PRORVnet). Right Ventricular Injury Increases Mortality in Patients With Acute Respiratory Distress Syndrome on Veno-Venous Extracorporeal Membrane Oxygenation: A Systematic Review and Meta-Analysis. ASAIO J. 2023 Jan 1;69(1):e14-e22. doi: 10.1097/MAT.0000000000001854. Epub 2022 Nov 13. PMID 36375040
- [Background] Dugar S, Sato R, Zochios V, Duggal A, Vallabhajosyula S; Protecting the Right Ventricle Network (PRORVnet). Defining Right Ventricular Dysfunction in Acute Respiratory Distress Syndrome. J Cardiothorac Vasc Anesth. 2022 Feb;36(2):632-634. doi: 10.1053/j.jvca.2021.09.001. Epub 2021 Sep 16. No abstract available. PMID 34583852
- [Result] Nasa P, Jain R, Juneja D. Delphi methodology in healthcare research: How to decide its appropriateness. World J Methodol. 2021 Jul 20;11(4):116-129. doi: 10.5662/wjm.v11.i4.116. eCollection 2021 Jul 20. PMID 34322364